CLINICAL TRIAL: NCT06665880
Title: The Changes of Genes, Proteins, and Metabolites in Patients with Drug-resistant Epilepsy
Brief Title: Genes, Proteins, and Metabolites in Drug-resistant Epilepsy (DRE) Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: Brain Tissues
Record Dates: First submitted 2024-08-05; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Drug Resistant Epilepsy; Traumatic Brain Injury Without Open Intracranial Wound
Keywords: Genomics; Proteomics; Metabolomics; Drug Resistant Epilepsy; Traumatic Brain Injury
MeSH Terms: conditions — Drug Resistant Epilepsy; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Epileptogenic and para-epileptogenic tissues from DRE patients and normal tissues from individuals with traumatic brain injury.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- DRE patients: Patients with drug-resistant epilepsy.
  Interventions: Other: Routine clinical treatment
- Traumatic Brain Injury: Individuals with traumatic brain injury.
  Interventions: Other: Routine clinical treatment

INTERVENTIONS:
Other: Routine clinical treatment — Routine clinical treatment is based on the latest international guidelines for DRE.

SUMMARY:
In patients with drug-resistant epilepsy (DRE), there may be changes at the genetic, proteomic, and metabolomic levels when comparing epileptic tissues from DRE to normal tissues in traumatic brain injury (TBI). These changes could help in understanding the pathophysiological mechanisms of epilepsy and in identifying new therapeutic targets.

DETAILED DESCRIPTION:
Genomical studies have identified changes in the expression of certain genes within epileptic tissues. These genes may be involved in pathways related to the balance of neuronal excitability and inhibition, synaptic transmission, and cell apoptosis.

Proteomic studies will reveal changes in the abundance and modifications of proteins in epileptic tissues. These could involve proteins related to the control of neuronal excitability and synaptic transmission, such as ion channels, neurotransmitter receptors, and synaptic proteins.

Metabolomic researches will reveal changes in metabolites within epileptic tissues. Epilepsy may lead to disruptions in metabolic pathways, affecting key processes such as energy metabolism, amino acid metabolism, and lipid metabolism.

Sample Size: There is no minimum or maximum, but is expected to be far less than 10.

In summary, patients with drug-resistant epilepsy might have changes in genes, proteomics, and metabolomics within epileptic tissues compared to normal tissue from TBI. Further research into these changes will deepen our understanding of the pathophysiology of epilepsy and guide the need for new treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

1. 14-60 years old, male or female, Han Chinese;
2. Drug-resistant epilepsy;
3. Required surgical implantation of SEEG electrodes.

Exclusion Criteria:

1. Progressive encephalopathy or progressive structural damage in the central nervous system;
2. Significant heart, liver, renal insufficiency, and other medical diseases;
3. Severe side effects from taking antiepileptic drugs at the time of enrollment and not inappropriate for SEEG;
4. Significant intellectual disability;
5. A history of alcohol and drug abuse;
6. Any contraindication to MRI.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with drug-resistant epilepsy.
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Single cell RNA sequencing | through study completion, an average of one year
  Cancerous and paracancerous tissues of patients will be subjected to10x Genomics single-cell RNA sequencing, Bulk RNA-seq and spatial transcriptome.

SECONDARY OUTCOMES:
Differentially expressed proteins | through study completion, an average of one year
  Discovering differentially expressed proteins (DEPs) and their roles in DRE patients, we will conduct 4D-DIA quantitative proteomics analysis.
The concentration of metabolites | through study completion, an average of one year
  Metabolites of cancerous and paracancerous tissues in patients will be subjected to LC-MS/MS, GC-MS and Desorption Electrospray Ionization - Imaging Mass Spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Guoguang Zhao, MD & PhD, Principal Investigator — Xuanwu Hospital, Beijing; Hongxing Wang, MD & PhD, Study Director — Xuanwu Hospital, Beijing; Yongzhi Shan, MD & PhD, Study Director — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No